Study Title: Project Insight: Feasibility of a Breast Cancer Screening Decision Support Tool

NCT#: NCT04741503

Date of Consent Document: 04/07/2021

FOR IRB USE ONLY
IRB ID #: 202101073
APPROVAL DATE: 04/07/21
RELEASED DATE: 04/08/21
EXPIRATION DATE: N/A

We invite you to participate in a research study being conducted by investigators from Washington University in St. Louis.

This is a research study conducted by Dr. Ashley Housten having to do with what women know and what they think about breast cancer screening. We are also asking women what they think about breast cancer screening informational materials. You may choose to participate or not. The National Institute on Minority Health and Health Disparities is funding this research study.

If you agree to participate, you will be volunteering to participate in the research study. As a voluntary participant, you will be asked to spend less than 30 minutes answering a questionnaire, reviewing informational materials, and finishing with a final questionnaire. We will be asking basic information about yourself, what you know and think about breast cancer screening, and your thoughts about breast cancer screening informational materials. The main risks to you if you participate are that the questions about sensitive information may make you feel uncomfortable. You are free to skip any questions that you prefer not to answer. If you do not want to participate, you can close the browser to exit the survey.

You may benefit from volunteering because you will learn about breast cancer screening. There is no cost to you and you will be compensated through Qualtrics for being a volunteer participant.

Approximately 234 people will take part in this study at Washington University.

There could be risks such as hacking, phishing, tracking cookies, breach of confidentiality or privacy, lack of appropriate security measures, leaving the computer unattended, or not having a password that prevents others from accessing the computer or mobile phone. In addition to these, there may be other unknown risks, or risks that we did not anticipate, associated with being in this study.

You will not benefit personally. However, we hope that others may benefit in the future from what we learn as a result of this study.

You will not have any costs for being in this research study.

To help protect your confidentiality, all data will be stored electronically under password protection in a secured server. Study-related computers will be under firewall protection and will maintain automated virus update mechanisms. Timely notification regarding relevant patches will be provided. In addition, all study staff annually sign a confidentiality statement attesting to their understanding of, and willingness to abide by, written policies on research ethics and confidentiality. Access to the data entry website will be password protected and restricted to personnel trained to use the system.

Any report or article that we write will not include information that can directly identify you.

FOR IRB USE ONLY
IRB ID #: 202101073
APPROVAL DATE: 04/07/21
RELEASED DATE: 04/08/21
EXPIRATION DATE: N/A

The journals that publish these reports or articles require that we share your information that was collected for this study with others to make sure the results of this study are correct and help develop new ideas for research. Your information will be shared in a way that cannot directly identify you.

Federal regulatory agencies and Washington University, including the Washington University Institutional Review Board (a committee that reviews and approves research studies) and the Human Research Protection Office may inspect and copy records pertaining to this research. If we write a report about this study we will do so in such a way that you cannot be identified.

The Siteman Cancer Center at Washington University School of Medicine and Barnes-Jewish Hospital is supported by funding from the National Cancer Institute (NCI). To meet NCI requirements, identifiable information about you relating to your participation in this study will be stored in a secure database at the Siteman Cancer Center. This database may be reviewed by Siteman Cancer Center personnel. All information will be securely and confidentially maintained.

To further protect your privacy, this research is covered by a Certificate of Confidentiality from the federal government. This means that the researchers can refuse to disclose information that may identify you in any legal or court proceeding or to anyone who is not connected with the research except if:

- there is a law that requires disclosure, such as to report child abuse and neglect, or harm to self or others;
- you give permission to disclose your information, including as described in this consent form; or
- it is used for other scientific research allowed by federal law.

You have the right to share your information or involvement in this study with anyone at any time. You may also give the research team permission to disclose your information to a third party or any other person not connected with the research.

Your participation in this study is completely voluntary. You may choose not to take part at all. If you decide to participate in the study you may stop participating at any time. Any data that was collected as part of this study will remain as part of the study records and cannot be removed. If you decide not to take part in the study or if you stop participating at any time, you won't be penalized or lose any benefits for which you otherwise qualify.

If you do not wish to participate in this study or want to end your participation in the study, you can close the browser to exit the survey.

We encourage you to ask questions. If you have any questions about the research study itself, please contact: Ashley Housten, OTD, MSCI, (314) 454-7958 or email <a href="mailto:ahousten@wustl.edu">ahousten@wustl.edu</a>. If you feel you have been harmed from being in the study, please contact: Ashley Housten, OTD, MSCI, (314) 454-7958. If you have questions, concerns, or

FOR IRB USE ONLY IRB ID #: 202101073 APPROVAL DATE: 04/07/21 RELEASED DATE: 04/08/21 EXPIRATION DATE: N/A

complaints about your rights as a research participant, please contact the Human Research Protection Office at 1-(800)-438-0445 or email hrpo@wustl.edu. General information about being a research participant can be found on the Human Research Protection Office web site, <a href="http://hrpo.wustl.edu">http://hrpo.wustl.edu</a>. To offer input about your experiences as a research participant or to speak to someone other than the research staff, call the Human Research Protection Office at the number above.

Thank you very much for your consideration of this research study.